CLINICAL TRIAL: NCT02843893
Title: Evaluation of Pupillary Distension Reflexes, as a Tool for the Monitoring of Analgesia for Patients in Intensive Care.
Acronym: PUPILLO REA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 38RC12.207
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Failure of Respiratory Function
Keywords: Pupillary; Reflexes; Analgesia; Sedation
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intubated and Mechanically Ventilated Patients (Other): Intubated and Mechanically Ventilated Patients receiving by continuous intravenous an hypnotic sedation (midazolam or propofol) associate with a morphine type drug (fentanyl, sufentanil, rémifentanil, or morphine) since at least 6 hours and for a predictable duration over 24 hours.
  Interventions: Device: Measure the minimum intensity of a painful stimulation

INTERVENTIONS:
Device: Measure the minimum intensity of a painful stimulation — With Neurolight device.

SUMMARY:
Sedation-analgesia is an important therapy for patients in resuscitation. It requires a surveillance, in order to avoid excessive or insufficient dosages of sedative or nonmorphinics, sources of side effects. Yet, means of surveillance are limited in resuscitation care : variations of blood pressure and heart rate are not very sensitive criterias. Clinical scales to measure the sedation and analgesia level were proposed for patients in resuscitation, including the Richmond (RASS) sedation scale and the behavioural pain scale (BPS). The study of pupillary dilatation's reflex (RDP) due to a nociceptive stimulation is a tool proposed for the monitoring of the analgesia peroperative for patients under general anaesthetic. Yet, there isn't any study that measured the analgesia threshold by pupillometry for patients in resuscitation receiving a sedation-analgesia.

The main goal of this study is to measure the minimum intensity of a painful stimulation (tetanus), leading to a 10% raise of RDP in a cohort of patients in resuscitation care receiving sedation-analgesia continuously.

DETAILED DESCRIPTION:
Secondary goals will be to bring this measures back to the pain score BPS and the pupillary diameter measured during a painful care (tracheal aspiration), as well as morphinics dosage.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and Mechanically Ventilated Patients receiving by continuous intravenous an hypnotic sedation (midazolam or propofol) associate with a morphine type drug (fentanyl, sufentanil, rémifentanil, or morphine) since at least 6 hours and for a predictable duration over 24 hours.
* Both gender
* Adult over 18 years

Exclusion Criteria:

* Neuromuscular pathology that does not allow the use of clinical scales in order to measure sedation-analgesia : tetraplegia, resuscitation neuromyopathy, curares.
* Intracranial hypertension (intracranial pressure over 20 mmHg) whatever the cause (traumatique, vasculaire, tumorale).
* Dysautonomia altering the pupillary dilatation's reflex (RDP) : old diabetes with diabetic retinopathy, multiple sclerosis, systemic amylose.
* Treatment in progress which may affect the pupillary dilatation's reflex (RDP) : antiemetic (droperidol, métoclopramide), alpha-2 agoniste (clonidine).
* Ocular pathology
* Opiate addiction
* Refusal by a patient
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Measure of pupillary dilatation's reflex (RDP) | 13 seconds
  Vidéopupillometer Neurolight®

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Payen, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Sauder P, Andreoletti M, Cambonie G, Capellier G, Feissel M, Gall O, Goldran-Toledano D, Kierzek G, Mateo J, Mentec H, Mion G, Rigaud JP, Seguin P. [Sedation and analgesia in intensive care (with the exception of new-born babies). French Society of Anesthesia and Resuscitation. French-speaking Resuscitation Society]. Ann Fr Anesth Reanim. 2008 Jul-Aug;27(7-8):541-51. doi: 10.1016/j.annfar.2008.04.021. Epub 2008 Jun 24. No abstract available. French. PMID 18579339
- [Background] Carrion MI, Ayuso D, Marcos M, Paz Robles M, de la Cal MA, Alia I, Esteban A. Accidental removal of endotracheal and nasogastric tubes and intravascular catheters. Crit Care Med. 2000 Jan;28(1):63-6. doi: 10.1097/00003246-200001000-00010. PMID 10667500
- [Background] Lorente L, Huidobro MS, Martin MM, Jimenez A, Mora ML. Accidental catheter removal in critically ill patients: a prospective and observational study. Crit Care. 2004 Aug;8(4):R229-33. doi: 10.1186/cc2874. Epub 2004 Jun 2. PMID 15312222
- [Background] The management of the agitated ICU patient. Crit Care Med. 2002 Jan;30(1 Suppl Management):S97-123; quiz S124-25. No abstract available. PMID 11852874
- [Background] Kollef MH, Levy NT, Ahrens TS, Schaiff R, Prentice D, Sherman G. The use of continuous i.v. sedation is associated with prolongation of mechanical ventilation. Chest. 1998 Aug;114(2):541-8. doi: 10.1378/chest.114.2.541. PMID 9726743
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Chanques G, Jaber S, Barbotte E, Verdier R, Henriette K, Lefrant JY, Eledjam JJ. [Validation of the french translated Richmond vigilance-agitation scale]. Ann Fr Anesth Reanim. 2006 Jul;25(7):696-701. doi: 10.1016/j.annfar.2006.02.017. Epub 2006 May 15. French. PMID 16698231
- [Background] Puntillo KA, Morris AB, Thompson CL, Stanik-Hutt J, White CA, Wild LR. Pain behaviors observed during six common procedures: results from Thunder Project II. Crit Care Med. 2004 Feb;32(2):421-7. doi: 10.1097/01.CCM.0000108875.35298.D2. PMID 14758158
- [Background] Payen JF, Bru O, Bosson JL, Lagrasta A, Novel E, Deschaux I, Lavagne P, Jacquot C. Assessing pain in critically ill sedated patients by using a behavioral pain scale. Crit Care Med. 2001 Dec;29(12):2258-63. doi: 10.1097/00003246-200112000-00004. PMID 11801819
- [Background] Yang LL, Niemann CU, Larson MD. Mechanism of pupillary reflex dilation in awake volunteers and in organ donors. Anesthesiology. 2003 Dec;99(6):1281-6. doi: 10.1097/00000542-200312000-00008. PMID 14639139
- [Background] Barvais L, Engelman E, Eba JM, Coussaert E, Cantraine F, Kenny GN. Effect site concentrations of remifentanil and pupil response to noxious stimulation. Br J Anaesth. 2003 Sep;91(3):347-52. doi: 10.1093/bja/aeg178. PMID 12925472
- [Background] Constant I, Nghe MC, Boudet L, Berniere J, Schrayer S, Seeman R, Murat I. Reflex pupillary dilatation in response to skin incision and alfentanil in children anaesthetized with sevoflurane: a more sensitive measure of noxious stimulation than the commonly used variables. Br J Anaesth. 2006 May;96(5):614-9. doi: 10.1093/bja/ael073. Epub 2006 Mar 24. PMID 16565227
- [Background] Larson MD, Sessler DI, Washington DE, Merrifield BR, Hynson JA, McGuire J. Pupillary response to noxious stimulation during isoflurane and propofol anesthesia. Anesth Analg. 1993 May;76(5):1072-8. doi: 10.1213/00000539-199305000-00028. PMID 8484510
- [Background] Jeanne M, Joulin O. [The 18th meeting of the Societe Francophone d'Informatique et de Monitorage en Anesthesie-Reanimation (Sfimar)]. Ann Fr Anesth Reanim. 2011 Oct;30(10):770-1. doi: 10.1016/j.annfar.2011.08.007. Epub 2011 Sep 23. No abstract available. French. PMID 21945009
- [Background] Larson MD, Talke PO. Effect of dexmedetomidine, an alpha2-adrenoceptor agonist, on human pupillary reflexes during general anaesthesia. Br J Clin Pharmacol. 2001 Jan;51(1):27-33. doi: 10.1046/j.1365-2125.2001.01311.x. PMID 11167662
- [Background] Li D, Miaskowski C, Burkhardt D, Puntillo K. Evaluations of physiologic reactivity and reflexive behaviors during noxious procedures in sedated critically ill patients. J Crit Care. 2009 Sep;24(3):472.e9-13. doi: 10.1016/j.jcrc.2008.07.005. Epub 2009 Jan 17. PMID 19327307